CLINICAL TRIAL: NCT01645800
Title: Effects of Lysozyme On Acute Exacerbation of Chronic Obstructive Pulmonary Disease : A Randomised Placebo-Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYS-002
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: COPD
Keywords: Lysozyme hydrochloride; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lysozyme hydrochloride (Experimental)
  Interventions: Drug: Lysozyme hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lysozyme hydrochloride — LYL 90mg capsule: Three times daily for 52 weeks.
  Arms: Lysozyme hydrochloride
Drug: Placebo — Matching Placebo capsule: Three times daily for 52 weeks.
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the effectiveness in preventing exacerbation of 52 weeks lysozyme administration in patients with COPD.

ELIGIBILITY:
Inclusion criteria;

* Patients were eligible for inclusion in the study if they were over 20 years of age and below 85 years of age, and had a smoking history, a diagnosis of COPD, a ratio of FEV1 to forced vital capacity(FVC) of less than 70%, and a documented history of at least one exacerbation leading to any treatment within the previous year.

Exclusion criteria;

* Patients with egg allergy
* Patients with domiciliary oxygen therapy
* Patients with pneumonia or pulmonary tuberculosis
* Patients with severe cardiovascular disorder,severe kidney disorder, severe hepatic disorder, severe hematological disorder.
* Patients with cancer.

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Acute exacerbation of COPD | 52 weeks

SECONDARY OUTCOMES:
Yearly reduction in FEV1 and QOL assessed by CAT | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yukinori Sakata, Study Director — Drug Fostering and evolution Coodination Department, Corporate Regulattory Compliance, Safety and Quality Assurance Headquaters, Eisai Co., Ltd., Japan
Locations (25):
- Japan (25):
  - Nishio, Aichi-ken
  - Noda, Chiba
  - Fukuoka, Fukuoka
  - Kasuga, Fukuoka
  - Kyoto-gun, Fukuoka
  - Yanagawa, Fukuoka
  - Mabashi, Gunma
  - Takasaki, Gunma
  - Kitahiroshima, Hokkaido
  - Sapporo, Hokkaido
  - Himeji, Hyōgo
  - Takamatsu, Kagawa-ken
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Nagaoka, Niigata
  - Ōita, Oita Prefecture
  - Okayama, Okyama
  - Osaka, Osaka
  - Suita, Osaka
  - Chuo-ku, Tokyo
  - Edogawa-ku, Tokyo
  - Higashikurume, Tokyo
  - Koto-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Yamagata, Yamagata